CLINICAL TRIAL: NCT00568191
Title: Reliability of Threshold Algorithm in Age-Related Macular Degeneration: Stratus Versus Cirrus OCT
Brief Title: Stratus Versus Cirrus OCT in AMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Prof Susanne Binder, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Other Study IDs: EK 06-007-VK1
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization
Keywords: Age-related macular degeneration; choroidal neovascularization; Stratus OCT; Cirrus OCT
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: retinal thickness program Stratus OCT software 4.0
- 2: retinal cube 200x200 program of Cirrus OCT

SUMMARY:
The Cirrus OCT provides due to the spectral domain technology a 2-fold resolution than Stratus OCT generated in a comparable amount of time. Due to this higher resolution the retinal surface and the retinal pigment epithelium can be identified more clearly, a significantly reduced number of algorithm failures is expected

ELIGIBILITY:
Inclusion Criteria:

* Age>55 years
* Age-related macular degeneration

Exclusion Criteria:

* Not consented patients

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 55 years of either sex presenting with age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Number of algorithm failures assessed by Stratus OCT versus Cirrus OCT in the horizontal central line | only 1 examination

SECONDARY OUTCOMES:
Number of algorrithm failures in Stratus versus Cirrus OCT assessed in the whole scan | 1 examination

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Krebs, Principal Investigator — Ludwig Boltzmann Institute of Retinology and Biomicroscopic Lasersurgery
Locations (1):
- Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Krebs I, Falkner-Radler C, Hagen S, Haas P, Brannath W, Lie S, Ansari-Shahrezaei S, Binder S. Quality of the threshold algorithm in age-related macular degeneration: Stratus versus Cirrus OCT. Invest Ophthalmol Vis Sci. 2009 Mar;50(3):995-1000. doi: 10.1167/iovs.08-2617. Epub 2008 Nov 21. PMID 19029035